CLINICAL TRIAL: NCT00345397
Title: Percutaneous Colostomy for Bowel Management in Spinal Cord Injury
Brief Title: A Colonic Tube to Improve Bowel Function in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4203-R
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Constipation; Fecal Incontinence; Spinal Cord Injury
Keywords: cecostomy; colonoscopy; colostomy; constipation; endoscopy, gastrointestinal; fecal incontinence; percutaneous; quality of life; spinal cord injury
MeSH Terms: conditions — Constipation; Fecal Incontinence; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects Receiving PEC Tube (Experimental): Percutaneous Endoscopic Colostomy Tube (PEC) Placement
  Interventions: Device: Percutaneous endoscopic colostomy (PEC) tube

INTERVENTIONS:
Device: Percutaneous endoscopic colostomy (PEC) tube — PEC placement for antegrade enemas uses commercially available PEG tubes

SUMMARY:
The investigators want to know if placing a tube through the skin and into the colon to flush out the colon is safe and effective in helping spinal cord Veterans with bowel management.

DETAILED DESCRIPTION:
1. Objectives: This Quality of Life (QoL) outcomes project studies the ability of Percutaneous Colostomy (PC) to clinically benefit Spinal Cord Injury (SCI) patients' bowel management and, thereby, their lives. This project runs under an umbrella Investigational Device Exemption (IDE). Specific objectives include:

   Safety: Monitor adverse events, especially for any evidence suggesting that use of Percutaneous Endoscopic Gastrostomy (PEG) devices (high risk device) for PC might pose an unreasonable risk.

   Efficacy: Prospectively evaluate the ability of a PEG device to successfully function as a PC; the ability of a PC to work in its clinically indicated application; the ability of the application to yield clinical benefits; and the ability of the clinical benefit to impact QoL. Technical Questions: Seek insights on the use of Fluoroscopy and Re-Colonoscopy in PC placement.
2. Research Design: In this 36-Month unblinded intervention trial, each SCI subject serves as his or her own control. Using a commercially available PEG tube, PC is placed colonoscopically, typically into the cecum. Technically, PC is directly analogous to PEG. Pre-and post-PC bowel function and QoL will be defined and compared. This will be the first rigorous prospective trial of endoscopic PC, especially for antegrade irrigation in SCI adults. This project is intended to be foundational, laying the groundwork for a variety of future studies.
3. Methodology: Subjects are drawn from the general SCI population at Zablocki Veterans Affairs Medical Center (VAMC). These patients have already been pre-screened for prevalence of bowel dysfunction, compliance, interest in research participation, and specific case finding. The investigators will mail a 7-Day Diary of bowel management to the 111 potential subjects that the investigators identified as having bowel management significantly impact their QoL. Successful completion of the 7-Day Diary will serve as a secondary compliance screen and define baseline bowel function. If the subject is interested in PC, additional evaluations, including psychological testing and an SCI-Specific, 20-question, QoL instrument will be undertaken pre-PC. Repeated measures at approximately 12 months will allow determination of physiological efficacy and impact on QoL. Additional characterization of each subject may also allow us to retrospectively define predictors of success related to bowel motility, clinical characteristics, psychosocial factors, etc.

   Underlying this Outcomes study is a standard Safety and Efficacy evaluation of the PC procedure, itself. Details of technical aspects of implantation, risk attenuation strategies, and data monitoring / reporting are outlined in cooperation with the FDA. This IDE covers 25 patients but only under the direct supervision of Drs. Otterson or Berger and only at the Zablocki VAMC.
4. Clinical Relationships: The potential clinical impact of PC is large. There are 45,000 SCI Veterans and 200,000 SCI patients across the country. If the sample is representative, 20% or more of these may benefit from PC. The secondary impact on healthcare costs, caregiver burden, and even employability is yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* SCI Veteran followed at Zablocki VAMC
* High quality of life impact of bowels on survey
* Ability to cooperate with data collection and follow-up requirements

Exclusion Criteria:

* Unstable clinical disease
* Untreatable co-morbidities affecting gut function
* Colonic disease or surgery that might impact safety of Percutaneous Colostomy tube placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Otterson, MD, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Receiving PEC Tube: All Enrolled Subjects receiving PEC Placement
Period: Overall Study
Arm/Group | Subjects Receiving PEC Tube
Started | 7
Completed | 6
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects Receiving Percutaneous Endoscopic Colostomy (PEC): Quality of Life (QOL) evaluation before and after device placement
Arm/Group | Subjects Receiving Percutaneous Endoscopic Colostomy (PEC)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Bowel QoL
Description: Spinal Cord Injury (SCI) -Specific, 20-Question QoL Instrument used a Visual Analog Scale (VAS) for each item.
  These were scored by measurement and recording 1-10 along the scale (1 being best, 10 being worst) An average of the scores for the 20-items was calculated for each subject before and after Percutaneous Endoscopic Colostomy (PEC) Tube placement.
  A Global SCI-QoL Score was also recorded using the same VAS. The difference between these Intake and Exit scores was used to define change in SCI-Specific Quality of Life.
Time Frame: Exit data collected 1 year(+/- 6 mo) after Intake data collection / PEC placement
Population: Subjects completing both Intake and Exit assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Global SCI-QoL Score in Subjects Receiving PEC Tube: Global SCI-QoL Score before and after device placement
- SCI-Specific QoL Evaluation in Subjects Receiving PEC Tube: SCI-Specific QoL evaluation before and after device placement
Arm/Group | Global SCI-QoL Score in Subjects Receiving PEC Tube | SCI-Specific QoL Evaluation in Subjects Receiving PEC Tube
Number analyzed (Participants) | 6 | 6
units on a scale | -4.17 (3.55) | -3.65 (1.263)

ADVERSE EVENTS:
Time Frame: Reporting includes the evaluation period of 6-18 months between Intake and Exit evaluations, as well as up to 24 month additional observation.
Groups:
- Subjects Receiving PEC Tube: QoL evaluation before and after device placement
Arm/Group | Subjects Receiving PEC Tube
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving PEC Tube (N=7)
Death, unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia death during follow-up period
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving PEC Tube (N=7)
Hyponatremia (Renal and urinary disorders) | 1 (1)
Fistula (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Difficulty in recruitment from a limited population reduced our intended enrollment and prolonged our study.

This also reduced our statistical significance and limited our conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No